CLINICAL TRIAL: NCT01820286
Title: Trial of a Positive Psychology Intervention to Reduce Suicide Risk in Patients With Mood Disorders
Brief Title: Positive Psychology for Mood Disorders
Acronym: PPBPAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Jeff C. Huffman, MD, Medical Director of Inpatient Psychiatric Unit, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2012P002294
Record Dates: First submitted 2013-03-25; First posted 2013-03-28 (Estimated); Last update posted 2017-09-05 (Actual); Status verified 2017-09

CONDITIONS: Bipolar Disorder; Depression
Keywords: Bipolar disorder; Depression; Positive psychology
MeSH Terms: conditions — Bipolar Disorder; Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Positive psychology intervention (Experimental): 4-week positive psychology intervention of 1 positive psychology exercise per week. Exercises will include 1) recalling 3 good events, 2) writing a letter of thankfulness, 3) using a personal strength, 4) envisioning a best possible future.
  Interventions: Behavioral: Positive psychology intervention
- Recollection intervention (Active Comparator): 4-week recollection intervention of 1 recollection exercise per week. Exercises will include recalling events related to 1) daily activities, 2) health, 3) social life, 4) morning and evening.
  Interventions: Behavioral: Recollection intervention

INTERVENTIONS:
Behavioral: Positive psychology intervention
  Arms: Positive psychology intervention
Behavioral: Recollection intervention
  Arms: Recollection intervention

SUMMARY:
The investigators are doing this study to see if "positive psychology" can help adults with depression or bipolar disorder.

Positive psychology involves exercises-short tasks-that try to increase good feelings and emotions, like optimism, happiness, personal strengths, and well-being. Positive psychology exercises might include imagining a bright future, being grateful for good events, forgiving others, and doing kind acts for others.

The investigators want to see if practicing positive psychology exercises after leaving the hospital can increase feelings of hope, optimism, and positive thinking. The investigators are asking you to take part in this research study because you are in the hospital for depression or bipolar disorder.

This research study will compare "positive psychology exercises" to "control condition exercises." During the study, you may take part in control condition exercises instead of positive psychology exercises.

ELIGIBILITY:
Inclusion Criteria:

* Patient admitted to Massachusetts General Hospital Inpatient Psychiatric Unit
* Age 18 and older
* Able to read and write in English
* Admission diagnosis of major depressive disorder or bipolar affective disorder (current depressive episode), confirmed using the Mini International Neuropsychiatric Interview and inpatient chart review

Exclusion Criteria:

* Psychotic symptoms, as assessed using the Mini International Neuropsychiatric Interview and inpatient chart review
* Cognitive disorder, assessed using a six-item cognitive screen developed for research
* Primary admission diagnosis of substance use disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2013-03; Primary Completion 2016-06-10 (Actual); Study Completion 2016-06-10 (Actual)

PRIMARY OUTCOMES:
Feasibility of positive psychology exercises | 8 weeks
  Feasibility will be measured by:
  1. Completion rate of exercises
  2. Ease of exercises (rated on a 5-point scale)
  3. Helpfulness of exercises (rated on a 5-point scale)

SECONDARY OUTCOMES:
Impact of positive psychology exercises on positive affect | 8 weeks
  Positive affect will be measured by:
  1. Optimism score on the Life Orientation Test-Revised (scores range from 3 to 30, with higher scores indicating higher levels of optimism)
  2. Gratitude score on the Gratitude Questionnaire-6 (scores range from 6 to 42, with higher scores indicating higher levels of gratitude)
  3. Positive emotion score on the Positive and Negative Affect Scale (scores range from 10 to 50, with higher scores indicating higher levels of positive emotion)
Impact of positive psychology exercises on negative affect | 8 weeks
  Negative affect will be measured by:
  1. Hopelessness scores on the Beck Hopelessness Scale (scores range from 0 to 20, with higher scores indicating higher levels of hopelessness).
  2. Suicidal ideation scores on the Concise Health Risk Tracking scale (scores range from 12 to 60, with higher scores indicating higher levels of suicidal ideation)
  3. Depression scores on the Quick Inventory of Depressive Symptomatology-Self Report (scores range from 0 to 27, with higher scores indicating higher levels of depression)

CONTACTS AND LOCATIONS:
Overall Officials: Jeff C Huffman, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States